CLINICAL TRIAL: NCT03350022
Title: Pilot Study on Sham Feeding in Post-operative Gastrointestinal Surgery Infants
Brief Title: Sham Feeding Post-operative Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Weems, MD, Associate Professor of Pediatrics, Le Bonheur Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-05475-FB
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Newborn Morbidity; Oral Aversion; Gastroschisis; Bowel Obstruction; Short Bowel Syndrome
MeSH Terms: conditions — Gastroschisis; Intestinal Obstruction; Short Bowel Syndrome | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sham Feeding (Experimental)
  Interventions: Procedure: Sham Feeding

INTERVENTIONS:
Procedure: Sham Feeding — Sham feeding will be offered to participants.
  Other Names: Observation

SUMMARY:
The purpose of this pilot study is to evaluate a feeding technique, sham feeding, to promote adequate oral skills in order to prevent oral aversion and/or poor oral skills due to the delay in oral feeds for surgical reasons. Sham feeding is intended for infants who are expected to have a prolonged course without normal enteral feeding by mouth.

DETAILED DESCRIPTION:
There is a lack of literature and research on which to base interventions that intend to preserve and develop oral and motor feeding skills in the post-operative patient population during the critical window of opportunity to establish proper oral skills. Due to the lack of positive oral feeding stimuli (i.e. prolonged airway management, nasogastric tubes, and airway and upper GI suctioning), these patients are at risk to develop oral aversions that may negatively impact long-term outcomes.

Parents in the neonatal intensive care unit (NICU) report feelings of stress and loss of control associated with medical interventions. When normal oral feeding is contraindicated, there may be impairment of parent-child bonding and mothers may be less dedicated to providing milk for the infant. Impaired bonding has been shown to affect the parent-child relationship and the child's development long after discharge.

Sham feeding has been shown to be safe and shorten time to oral feeding in infants with esophageal atresia with delayed esophageal repair. Anecdotal evidence from Le Bonheur suggests that sham feeding in post-operative gastroschisis patients improves parental satisfaction and engagement.

There is no literature to describe the use of sham feeding in neonates other than those with esophageal atresia. Anecdotal reports from our institution and others institutions suggests that it increases parental engagement and improves parental satisfaction among patients with other bowel pathology.

This is a cohort study with historical controls within a single level IV NICU. Participants will be offered sham feeding by breast or bottle and observed.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates at least 34 weeks post-menstrual age who have a history of gastrointestinal surgery, require no respiratory support more than 2 lpm by nasal cannula, and have an anticipated prolonged course with contraindication to normal oral or enteral feeding. They must have a diagnosis of gastroschisis awaiting return of bowel function, bowel atresia or other obstruction with anticipated feeding contraindication longer than 30 days, or short bowel syndrome intolerant of full intermittent oral feeding.
2. Mothers of enrolled neonates

Exclusion Criteria:

1. Lack of consent or parental consent.
2. Contraindication to sham feeding as determined by the responsible medical provider.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Time to full feeds | 1 year
  Time to full oral feeds after resolution of feeding contraindications

SECONDARY OUTCOMES:
Growth | 1 year
  Infant growth parameters
Duration of breast feeding | 1 year
  Duration of breast feeding or pumping of mother's milk
Maternal satisfaction | 1 year
  Maternal satisfaction survey after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weems, MD, Principal Investigator — University of Tennessee
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No